CLINICAL TRIAL: NCT02314650
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Propofol Consumption During General Anesthesia
Brief Title: TEAS to Reduce Propofol Consumption During General Anesthesia
Acronym: TOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Dr, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-A-2014-6-25-01
Record Dates: First submitted 2014-12-07; First posted 2014-12-11 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Transcutaneous acupoint stimulation (Experimental): Electrical stimulation was given through electrodes attached to skin at Ximen and Shenmen acupoint during anesthesia
  Interventions: Other: acupoint stimulation; Other: electrodes attached
- Non-acupoint stimulation (Placebo Comparator): Electrical stimulation was given through electrodes attached to skin at shoulder (non-acupoint) during anesthesia
  Interventions: Other: non-acupoint stimulation; Other: electrodes attached
- Control (Sham Comparator): patients were with electrodes attached but no stimulation was given
  Interventions: Other: electrodes attached

INTERVENTIONS:
Other: acupoint stimulation — stimulation was given at acupoints
  Arms: Transcutaneous acupoint stimulation
Other: non-acupoint stimulation — stimulation was given at non-acupoints
  Arms: Non-acupoint stimulation
Other: electrodes attached — electrode were attached to skin

SUMMARY:
The study is aimed at whether transcutaneous electrical acupoint stimulation (TEAS) during general anesthesia could reduce the need for propofol in patients undergoing minor surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing minor surgeries including laparoscopic surgery and breast surgery under general anesthesia
* Patients with written informed consent

Exclusion Criteria:

* Patients with difficulty to communicate,including psychiatric disorder and Alzheimer's disease
* Patients with drug abuse
* Patients with disease of central nervous system
* Patients with renal or hepatic dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
propofol consumption | from induction to the end of surgery,at an average of 1 hour

SECONDARY OUTCOMES:
time to awake | from end of propofol infusion to open eyes to verbal command,at an average of 30 minutes
time to extubation | from end of propofol infusion to open eyes to verbal command,at an average of 30 minutes
effect site concentration of propofol at awake | from end of propofol infusion to open eyes to verbal command,at an average of 30 minutes
highest sedation score during stay at postanesthesia care unit | from end of surgery to discharge from post anesthesia care unit, at an average of 1 hour
nausea and vomiting during stay at postanesthesia care unit | 30min after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong LU, PhD, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Result] Fassoulaki A, Paraskeva A, Patris K, Pourgiezi T, Kostopanagiotou G. Pressure applied on the extra 1 acupuncture point reduces bispectral index values and stress in volunteers. Anesth Analg. 2003 Mar;96(3):885-890. doi: 10.1213/01.ANE.0000048713.41657.D3. PMID 12598279
- [Result] Nayak S, Wenstone R, Jones A, Nolan J, Strong A, Carson J. Surface electrostimulation of acupuncture points for sedation of critically ill patients in the intensive care unit--a pilot study. Acupunct Med. 2008 Mar;26(1):1-7. doi: 10.1136/aim.26.1.1. PMID 18356793